CLINICAL TRIAL: NCT06353607
Title: Genetic Architecture of Acute Aortic Syndromes and Aortic Aneurysm.
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-02267; kt23Berdajs
Record Dates: First submitted 2024-04-02; First posted 2024-04-09 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Acute Aortic Dissection; Thoracic Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to explore the genetic information associated with the development of TAA and aAD in individuals without history or syndromic features (Marfan syndrome, Ehlers-Danlos syndrome, Turner syndrome etc.) for aortic disease. For this purpose, whole genome sequencing will be performed in patients with documented aortic aneurysm or/and aortic dissection.

DETAILED DESCRIPTION:
Acute aortic dissection (aAD) is a life-threatening condition, associated with increased morbidity and mortality. The incidence of aAD has been estimated to occur at a rate of 6-7 cases per 100.000 persons per year and is associated with high mortality. With the increasing availability of computed tomography scan (CT) in emergency settings, the diagnosis of aAD was increasing in past decades, increasing up to 17 cases per 100.000 persons per year. Acute aortic event is associated with a high mortality rate ranging from 26% in surgically treated patients to 58% in medically treated patients.

Thoracic aortic aneurysm (TAA) is a well-established risk factor for aAD but it is not a prerequisite. Recent evidence suggests that almost 90% of aAD's occur mostly in younger patients with aortic dimensions of <5.5 cm and only 5% of patients with diagnosed TAA are symptomatic prior to dissection or rupture.

The majority of aAD patients are misdiagnosed, which puts them at a higher risk of death. Timely diagnosis and surgical management of patients with TAA prior to aAD reduces the risk of complications and death. Therefore, there is an unmet need for better and more refined risk prediction tools to identify high-risk patients with TAA, who may benefit from early screening and tuned surgical intervention.

Previous studies found that more than 20% of patients with TAA report a positive family history, and the genetics of thoracic aortic aneurysm and dissection has been extensively investigated as a potential tool for both diagnosis and risk stratification.

Traditionally, TAA is divided into syndromic-with other organ system abnormalities other than the aorta-and non-syndromic-with no systemic abnormalities present. Several monogenic causes for syndromic TAA are well described, such as Marfan syndrome (MFS), Loeys-Dietz syndrome (LDS), and Ehlers-Danlos syndrome (EDS). However, the non-syndromic TAA and aAD are more prevalent, and identifying these patients can be challenging. Some evidence exist that mutations of genes observed in syndromic patients may be involved in TAA and aAD in non-syndromic patients. The fact that approximately 20% of non-syndromic TAA patients have at least one affected family member indicates that TAA could be a heritable disease and there might be a genetic link in non-syndromic patients.

Given the inherent challenges in the diagnosis of the TAA as a precursor of aAD in non-syndromic patients, there is a clinical need for the development of an accurate risk prediction tools. To address the mentioned clinically relevant question, in an observational cohort study of patients with aortic disease a molecular genetic investigation will be conducted to investigate the genetic architecture of TAA and individuals at high risk for aAD, and to use this information to propose patient specific risk assessment and individually tailored management and therapy. This data will be coupled to the routinely collected standard clinical and imaging data including computed tomography angiography (CTA), perioperative transesophageal echocardiogram (TEE) and transthoracic echocardiogram (TTE) with the aim to further refine risk stratification in aAD/TAA patients.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients > 18 years who underwent surgery for aAD or TAA intervention at the University Hospital Basel, starting in 2015.
* All patients who will undergo surgery for aAD or TAA at the University Hospital Basel, beginning in 2024.

Exclusion Criteria:

* Patients will be excluded if they are not able or not willing to provide informed consent.
* Patients with diagnosed heritable vascular disorders, such as Marfan syndrome, Turner Syndrome, Loeyes Dietz and Ehlers-Danlos syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with surgical aAD or TAA intervention performed at the Unversity Hospital Basel between 2015 and 2028.
Sampling Method: Non-Probability Sample
Enrollment: 730 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the association between the prevalence of TAA and/or aAD in variants with genes associated with thoracic aortic disease. | Baseline to last follow-up visit (up to 4 years)
  Assessment of the association between the prevalence of TAA and/or aAD in variants with genes associated with thoracic aortic disease.

SECONDARY OUTCOMES:
Investigate the genetic landscape of aortic specimens retrieved from surgical intervention tissues, and relate the genetic profile to cell molecular pathology. | Baseline to last follow-up visit (up to 4 years)
  Investigate the genetic landscape of aortic specimens retrieved from surgical intervention tissues, and relate the genetic profile to cell molecular pathology.
To assess the association between the aortic segment dimension (in CT scan and TEE images), tissue pathology and gene variants to determine the images predictive factors for TAA and/or aAD. | Baseline to last follow-up visit (up to 4 years)
  To assess the association between the aortic segment dimension (in CT scan and TEE images), tissue pathology and gene variants to determine the images predictive factors for TAA and/or aAD.
To establish a risk prediction model for aAD and TAA based on genetic, clinical, and imaging endpoints. | Baseline to last follow-up visit (up to 4 years)
  To establish a risk prediction model for aAD and TAA based on genetic, clinical, and imaging endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Berdajs, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided